CLINICAL TRIAL: NCT03620760
Title: A Prospective, Randomised, Open-labeled, Parallel Group Study to Assess the Efficacy and Safety of Low Dose Ticagrelor Compared With Standard Dose Ticagrelor in Patients With Unstable Angina Pectoris After Drug Eluting Stent Implantation
Brief Title: Efficacy and Safety of Low Dose Ticagrelor in Patients With Unstable Angina Pectoris After Coronary Stent Implantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaofan Wu (Other)
Responsible Party: Sponsor-Investigator, Xiaofan Wu, Chief Physician, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-2-1064
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Unstable Angina Pectoris; Coronary Stent Implantation
Keywords: Unstable Angina; Stent; Ticagrelor; Platelet aggregation; Percutaneous Coronary Intervention; Coronary Artery Disease; Major Adverse Cardiovascular and Cerebrovascular Events; Bleeding Events
MeSH Terms: conditions — Angina, Unstable; Coronary Artery Disease | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Intervention Model Description: Eligible patients were randomly assigned in a 1:1 ratio to receive ticagrelor 90 mg twice daily plus aspirin 100mg once daily or ticagrelor 45 mg twice daily plus aspirin 100mg once daily.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower dose ticagrelor (Experimental): Subjects will be treated with ticagrelor 45 mg twice daily in combination with aspirin 100mg once daily.
  Interventions: Drug: Ticagrelor 45 mg; Drug: Aspirin
- Standard dose ticagrelor (Active Comparator): Subjects will be treated with ticagrelor 90 mg twice daily in combination with aspirin 100mg once daily.
  Interventions: Drug: Ticagrelor 90 mg; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor 90 mg — Ticagrelor (AZD6140) 90 mg twice daily dose
  Other Names: AZD6140
  Arms: Standard dose ticagrelor
Drug: Ticagrelor 45 mg — Ticagrelor (AZD6140) 45 mg twice daily dose
  Other Names: AZD6140
  Arms: Lower dose ticagrelor
Drug: Aspirin — Aspirin 100 mg once daily dose

SUMMARY:
The study is to evaluate efficacy and safety of low dose of ticagrelor therapy for Chinese unstable angina patients treated with non-urgent coronary stent implantation, to examine whether lower dose ticagrelor (45 mg twice-daily) is not inferior to standard dose (90 mg twice-daily) for the prevention of major adverse cardiovascular and cerebrovascular events, as well as will reduce the incidence of bleeding during long-term treatment.

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, parallel-group trial designed to evaluate the efficacy and safety of low dose ticagrelor on a background of aspirin for patients treated with non-urgent coronary stent implantation. 2036 subjects will be enrolled. All patients will receive treatment with aspirin and a P2Y12 inhibitor for 3 months after the index procedure. At 3 months, eligible patients were then randomly assigned in a 1:1 ratio to receive a standard dose ticagrelor 90 mg bid or a lower dose ticagrelor 45 mg bid in addition to aspirin 100mg. The primary efficacy end points are the event rate of the composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis, coronary revascularization and stroke at 24 months. The primary safety end point is the incidence of PLATO major bleeding at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients admission for coronary artery disease treatment with non-emergency percutaneous intervention with stent deployment
* 18 years≤age≤80 years
* Patients understands the study requirements and the treatment procedures and provided informed consent before the procedure

Exclusion Criteria:

* Allergy or intolerance to ticagrelor or aspirin
* Need for oral anticoagulation therapy
* Concomitant oral or intravenous therapy with strong inhibitors of Cytochrome P450, family 3, subfamily A (CYP3A), Substrates of CYP3A with narrow therapeutic indices or strong inducers of CYP3A
* Active bleeding, previous history of intracranial hemorrhage, gastrointestinal hemorrhage in the past 6 months and major operation within 30 days
* High risk of bradyarrhythmias
* Severe liver dysfunction and abnormal renal function
* Patient is a woman who is pregnant or nursing
* Unable or unwilling to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2036 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular and cerebrovascular events (MACCEs) and major bleeding event | Randomization up to 24 months
  Participants with death from vascular causes, non-fatal myocardial infarction, stent thrombosis, coronary revascularization and stroke. Intention to treat (ITT) analysis of whole population. Events were adjudicated by an endpoint committee.
  Participants with PLATO major bleeding event including fatal bleeding, intracranial bleeding, intrapericardial bleeding with cardiac tamponade, hypovolemic shock or severe hypotension due to bleeding and requiring pressures or surgery, a decline in the hemoglobin level of 5.0 g per deciliter or more, or the need for transfusion of at least. Events were adjudicated by an endpoint committee.

SECONDARY OUTCOMES:
Any event from the composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis, coronary revascularization and stroke | Randomization up to 24 months
  Participants with any event from the composite of cardiovascular death, non-fatal MI, stent thrombosis, coronary revascularization and stroke. ITT analysis of intent for invasive management population. Events were adjudicated by an endpoint committee.
All cause death | Randomization up to 24 months
  Participants with all cause death. ITT analysis of whole population. Events were adjudicated by an endpoint committee.
PLATO-defined any bleeding event | Randomization up to 24 months
  Participants with any other bleeding events (minor bleeding or minimal bleeding) as defined by the PLATO. Events were adjudicated by an endpoint committee.

OTHER OUTCOMES:
PLATO-defined any minor bleeding event | Randomization up to 24 months
  To compare two intensities of ticagrelor therapy on minor bleeding event as any bleeding requiring medical intervention but not meeting the criteria for major bleeding. Events were adjudicated by an endpoint committee.
PLATO-defined any minimal bleeding event | Randomization up to 24 months
  To compare two intensities of ticagrelor therapy on minimal bleeding event as all other bleeding (eg, bruising, bleeding gums, oozing from injection site) not requiring intervention or treatment. Events were adjudicated by an endpoint committee.
Other adverse events | Randomization up to 24 months
  To compare two intensities of ticagrelor therapy on other adverse events including dyspnea or bradyarrhythmia. Events were adjudicated by an endpoint committee.
Experiment examination | Randomization up to 24 months
  To compare two intensities of ticagrelor therapy on increase of serum uric acid or creatinine. Events were adjudicated by an endpoint committee.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Wu, Study Director — Beijing Anzhen Hospital
Locations (1):
- Xiaofan Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No